CLINICAL TRIAL: NCT06511115
Title: New Technologies for Improving Physical, Mental, and Cognitive Health in Older Adults
Brief Title: New Technologies for Enhancing Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJA.
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Older People

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Technologies Group (Experimental): Participants assigned to the experimental group will engage in an exercise program using technologies, including the Nintendo Wii, over a 12-week period, with a frequency of 3 sessions per week, each lasting 45 minutes.
  Interventions: Other: Experimental Group
- Control Group (No Intervention): This group will not undergo the physical exercise intervention but will receive general recommendations for comprehensive health care. These include information about the benefits of physical exercise and tips for managing physical and mental health. The control group (CG) will undergo all the proposed physical and mental tests at the beginning of the study and again after 12 weeks. Additionally, during the study period, they will be monitored for changes in physical activity levels, as well as nutritional changes, sleep habits, and stress levels.

INTERVENTIONS:
Other: Experimental Group — Each session will be divided into three clearly differentiated parts:
  i) A 5-minute warm-up consisting of a series of gentle, low-intensity exercises designed to gradually prepare the muscles and joints of older adults for the main exercise. This portion will include flexibility and stretching movements, as well as joint mobility exercises; ii) 35 minutes dedicated to the main section of the intervention using the Nintendo Wii to promote physical, mental, and cognitive activity; iii) 5 minutes for relaxation techniques that incorporate flexibility exercises and stretches.
  Each session will be led by a qualified and experienced professional. No incidents of injuries or negative effects were reported during the intervention period. Throughout the 12-week intervention, participants will be periodically followed up by phone to inquire about their physical activity habits.
  Arms: New Technologies Group

SUMMARY:
New technologies, such as mobile apps, health monitoring devices, interactive video games, and telemedicine platforms, have become invaluable for improving the physical, mental, and cognitive health of older adults. They help maintain flexibility, strengthen muscles, improve balance and posture, alleviate chronic pain, enhance sleep quality, and reduce stress and anxiety. Tools like the Nintendo Wii promote physical activity, improve coordination, and offer social interaction. Overall, these technologies support better mental health, emotional well-being, and independence, contributing to a higher quality of life for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older.
* Present physical autonomy to participate in the technological and physical activities required by the study.
* Present current affiliation to the social health security system.
* Sign the informed consent.
* Understand the instructions, programs and technological protocols of this project.
* Complete more than 90% of the intervention with technology and exercise.

Exclusion Criteria:

* Present medical contraindications for performing physical tests or using technologies.
* Present diseases that limit cognitive performance and physical activity.
* Present vestibular diseases.
* Present rheumatological diseases that can be exacerbated by the use of technologies or stress articulate.
* Refusing to sign the informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Balance and gait | Up to twelve weeks
  Tinetti. Completion time: 8-10 minutes. While walking behind the patient, the evaluator asks them to respond to the questions from the gait subscale. To answer the balance subscale, the interviewer stands next to the patient. A higher score indicates better functioning. The maximum score for the gait subscale is 12, and for the balance subscale, it is 16. The sum of both scores is used to assess the risk of falls. A higher score indicates a lower risk. A score of less than 19 signifies a high risk of falls.
Chair sit and reach test | Up to twelve weeks
  The test measures low back and hamstring flexibility. Sitting on a chair against a wall, one foot stays flat on the floor. Extend the other leg forward with knee straight, heel down, and ankle bent at 90°. Stack hands with middle fingers aligned. Inhale, then exhale while reaching toward toes without bouncing or pain. Keep back straight and head up, holding the stretch for 2 seconds. Measure distance between fingertips and toes: zero if touching, negative if not touching, positive if overlapping. Record to nearest 1/2 inch or 1 cm, noting which leg was used.
Back scratch test | Up to twelve weeks
  The shoulder range of motion test is conducted standing. Place one hand behind the head and over the shoulder, reaching down the middle of your back with palm touching your body and fingers pointing downwards. The other hand goes behind your back, palm out and fingers up, aiming to touch or overlap the middle fingers of both hands. An assistant aligns fingers and measures the distance between their tips. Score zero if fingertips touch, negative if not touching, positive if overlapping. Perform two practice attempts and two test attempts, stopping if pain occurs. Record the best score to the nearest centimeter or half inch for assessment.
30 second chair stand test | Up to twelve weeks
  Evaluates lower extremity strength. To perform the chair stand test: Use a chair with a 44 cm high seat and no armrests, secured against a wall. Ensure consistency by using the same chair for future tests. Participants should wear comfortable sports or walking shoes. Sit with feet flat on the floor, shoulder-width apart, knees slightly bent over 90 degrees, and heels closer to the chair than knees. Cross arms over chest. Start the stopwatch and instruct the participant to stand up fully and sit down, counting each cycle as one repetition within 30 seconds. If the 30-second mark aligns mid-action (standing up or sitting down), count it as a full repetition. Participants can rest during the test, but timing continues until 30 seconds elapsed.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No